CLINICAL TRIAL: NCT04522739
Title: Spironolactone Safety in African Americans With Mild Cognitive Impairment and Early Dementia
Acronym: STAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Principal Investigator, Antoine Trammell, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00000124
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Experimental): Participants with mild cognitive impairment or early Alzheimer's Disease who are randomized to receive spironolactone for 12 months.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Participants with mild cognitive impairment or early Alzheimer's Disease who are randomized to receive a placebo to match spironolactone for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Study participants will receive a 25 mg dose of spironolactone. Participants will take one capsule by mouth per day for 12 months.
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — A placebo to match spironolactone will be taken orally once per day for 12 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether a blood pressure medication, spironolactone, can be tolerated by older African American adults that have memory and thinking problems, also called mild cognitive impairment (MCI). This study will also investigate the effect of spironolactone on memory and thinking abilities as measured by performance on cognitive tests, which are tests that measure memory and thinking skills. Participants will take spironolactone or a placebo for one year and will have 4 to 5 study visits during the study period.

DETAILED DESCRIPTION:
In 2018, 5.5 million older adults in the United States were diagnosed with Alzheimer's disease, and it is predicted that 15 million people will be diagnosed with dementia, including Alzheimer's disease by 2060. Older African Americans adults are more likely to be diagnosed with Alzheimer's disease as compared to Whites. Research search studies on high blood pressure show that African Americans have higher levels of the hormone aldosterone that can be involved with regulation of blood pressure and blood vessels. Research studies also show that changes in blood vessels in the brain from higher aldosterone levels are related to changes in thinking skills and memory (cognition). Spironolactone is a drug that blocks aldosterone and has been used to treat high blood pressure for 60 years. More recently, this drug has shown to have the potential to decrease declines in thinking skills and memory.

Spironolactone is widely used in clinical practice and is well-tolerated by younger and older persons. As such, this study is designed to learn how a small group of older African American adults with mild cognitive impairment will tolerate the drug. Persons who are eligible for the study and agree to participate will receive spironolactone or a placebo and be monitored for drug side effects for one year.

During the study, the researchers will monitor changes in thinking and memory and blood vessel stiffness, in addition to side effects that may be related to the drug. Study tests include questionnaires that evaluate thinking skills and memory, and an ultrasound that measures the stiffness of blood vessels in the neck which deliver blood to the brain. The thinking and memory tests and ultrasound will be performed at the beginning of the study, then repeated at the end of the study.

The results of this study can justify a larger size study of spironolactone in older African Americans with mild cognitive impairment. The study has the potential to identify a new use for a well-known drug that is safe and widely used in current clinical practice. Further, the results from this study can address a racial difference in Alzheimer's disease and preserve the health of the brain as people age.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Willingness to comply with all study procedures and availability for the duration of the study
* Self-identified African American
* Blood pressure (BP) and hypertension criteria: normotensive and hypertensive participants will be eligible

  * Normotensive criteria: BP 110-140/40-90 mmHg and not receiving any treatment for hypertension
  * Hypertensive criteria: only controlled hypertensives will be eligible with BP range as in the normotensive criteria of 110-140/40-90 mmHg
* MCI defined as:

  * Abnormal memory function per the Logical Memory subscale (Delayed Paragraph Recall, Paragraph A only) from the Wechsler Memory Scale-Revised (the maximum score is 25):

    * Score <11 for 16 or more years of education
    * Score <9 for 8-15 years of education
    * Score <6 for <7 years of education
    * Montreal Cognitive Assessment (MoCA) score 13-25
    * Preserved general functional performance per Functional Assessment Questionnaire (FAQ)<9

Exclusion Criteria:

* History of stroke in the previous three years
* MoCA<13 or the inability to follow instructions to perform cognitive testing
* Inability to participate in the study procedures: cognitive tests (communication limitations from language or other factors)
* Active medical problem/symptom that interferes with the study procedures, e.g., chest pain, shortness of breath, or abdominal pain
* Deemed ineligible by study investigators due to safety issues or non-compliance
* History of the inability to tolerate treatment with an aldosterone antagonist
* Hypertension

  * Uncontrolled defined as a BP > 140/90 mmHg
  * Current therapy with RAAS modulating medications, i.e., angiotensin II receptor blocker (ARB), angiotensin converting enzyme inhibitor (ACEi), renin inhibitor, or aldosterone antagonist such as eplerenone (Inspra) due to the risk of hyperkalemia and the interference with the renin angiotensin aldosterone system (RAAS) system
* Renal disease (baseline creatinine > 2.0 mg/dL)
* Hyperkalemia (K+ > 5.5 milliequivalent (mEq)/dL)
* Other neurological or psychiatric conditions that could impact cognition, e.g., Parkinson's disease and related movement disorders, multiple sclerosis, epilepsy, or schizophrenia, untreated major depressive disorder, and other psychotic disorders
* Abnormal thyroid stimulating hormone (TSH) (>10 milliunits (mU)/L) or vitamin B12 (<250 pg/mL) as they can impact cognitive function. If the potential participant's TSH and/or vitamin B12 levels are abnormal, then the PI may enroll that person if it is thought the lab abnormalities are unrelated and do not affect cognitive function
* Active medical or psychiatric disease, which in the judgment of the study investigators affects participant safety or the scientific integrity of the study
* Uncontrolled congestive heart failure reflected by poor exercise tolerance and shortness of breath
* Women of childbearing potential, i.e., non-menopausal
* When potential participants are not capable of providing informed consent due to their cognitive impairment and a study partner/legally authorized representative (LAR) is not available to sign consent forms on their behalf

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Count of Adverse Events | Year 1
  The safely of the study treatment will be assessed with the number of adverse events experienced in each study arm.
Attrition rate | Year 1
  The tolerability of the study treatment will be assessed by the attrition rate of participants in each study arm.

SECONDARY OUTCOMES:
Change in Trail Making Test Part A Score | Baseline, Month 6, Month 12
  In Part A of the Trail Making Test (TMT) participants are presented with a sheet of paper with 25 circles numbered 1 through 25. Participants are asked to draw lines connecting the circles in ascending order of the numbers. The task is scored as the amount of time it takes in seconds for the circles to be correctly connected. The average time to complete the task is 29 seconds. Times greater than 78 seconds indicate cognitive impairment.
Change in Trail Making Test Part B Score | Baseline, Month 6, Month 12
  Part B of the Trail Making Test (TMT) includes a sheet of paper with circles with numbers (1-13) and letters (A-L). Participants are asked to draw lines connecting the circles in ascending order of the numbers and letters, alternating between numbers and letters. The task is scored as the amount of time it takes in seconds for the circles to be correctly connected. The average time to complete the task is 75 seconds. Times greater than 273 seconds indicate cognitive impairment.
Change in Hopkins Verbal Learning Test-Revised (HVLT-R) Total Recall Score | Baseline, Month 6, Month 12
  In the HVLT-R recall task, there are three trials where participants hear 12 words which they are asked to recall. The Total Recall score is the sum of correct responses over the three trials. Total scores range from 0 to 36 where higher scores indicate better recall.
Change in Hopkins Verbal Learning Test-Revised (HVLT-R) Delayed Recall Score | Baseline, Month 6, Month 12
  In the HVLT-R delayed recall task, participants hear 12 words and are asked to recall the words after waiting 20-25 minutes. The score is the sum of correctly recalled words and the score ranges from 0 to 12, where higher values indicate better delayed recall.
Change in Hopkins Verbal Learning Test-Revised (HVLT-R) Recognition Discrimination Index Score | Baseline, Month 6, Month 12
  In the HVLT-R recognition task, participants hear 24 words (half of which they have heard before) and are asked each each word has been previously presented. The recognition discrimination is calculated as the number of true positives minus the number of false positives during the recognition task. Index scores can range from -12 to 12 with higher scores indicating better recognition discrimination.
Change in Digit Span Test Score | Baseline, Month 6, Month 12
  The Digit Span test being used is a subtest of the Wechsler Adult Intelligence Scale - Third Edition (WAIS-III) and assesses immediate memory and attention. Participants are asked to repeat strings of numbers forwards and backwards. The score is the number of digits that are repeated correctly. Higher scores indicate improved memory and attention.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Trammell, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory Clinic at Executive Park, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared.
Supporting Information: Study Protocol
Time Frame: The data will become available beginning 36 months and ending three years following article publication.
Access Criteria: The data will be shared with researchers who provide a methodically sound proposal in order to achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in Emory University's data warehouse but without investigator support other than deposited metadata. Proposals should be directed to antoine.trammell@emory.edu. The requestors will need to sign a data access agreement to gain access to the data.